CLINICAL TRIAL: NCT01491594
Title: A Phase I/II Open-label Study of Eltrombopag for the Prevention of Chemotherapy Induced Thrombocytopenia (CIT) in Subjects With Advanced Soft Tissue and Bone Sarcomas Receiving Gemcitabine and Docetaxel Chemotherapy
Brief Title: Eltrombopag for the Prevention of Chemotherapy Induced Thrombocytopenia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to accrue subjects to the study.
Sponsor: Duke University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00032798
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2013-04

CONDITIONS: Sarcoma, Soft Tissue; Osteosarcoma; Neoplasms, Connective and Soft Tissue
Keywords: Metastatic sarcoma; Bone sarcoma
MeSH Terms: conditions — Sarcoma; Osteosarcoma; Neoplasms, Connective and Soft Tissue; Bone Neoplasms | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag is taken by mouth daily beginning 5 days before the start of each chemotherapy cycle for 10 days. In the phase 1 part of the study the dose will be 100, 150, 225, or 300 mg.
  Other Names: Promacta

SUMMARY:
The purpose of this study is to study the effect of eltrombopag on chemotherapy induced thrombocytopenia. Thrombocytopenia is when there is a low number of platelets in the blood. Sometimes, thrombocytopenia occurs as a side effect of chemotherapy treatments.

DETAILED DESCRIPTION:
The combination chemotherapy regimen of gemcitabine and docetaxel has become an increasingly used treatment choice for subjects with advanced sarcomas. The regimen has shown activity in first and second line for subjects with metastatic uterine leiomyosarcoma, relapsed/refractory pediatric sarcomas, and improved progression-free survival and overall survival in persons with metastatic sarcoma when compared to gemcitabine alone. The regimen has additionally been recognized as a treatment option for subjects with advanced sarcoma.

Chemotherapy-induced toxicity in the blood such as low platelet level is a common and often therapy-limiting side effect of treatment.

There are two phases in this study. The purpose of the Phase I study is to determine the recommended dose of eltrombopag. The purpose of the Phase II study is to determine the safety, tolerability, and efficacy (how well the drug works) of eltrombopag in subjects who are receiving gemcitabine and docetaxel chemotherapy.

Eltrombopag (Promacta) is an FDA approved drug for the treatment of chronic idiopathic thrombocytopenic purpura (ITP)- a condition of having an abnormally low platelet count. Eltrombopag is now being further investigated for other thrombocytopenic (low platelet)disorders.

Participants will take the assigned dose of eltrombopag once a day starting five days before each cycle of chemotherapy and for 5 days after chemotherapy. Eltrombopag is not taken on the day of chemotherapy. Eltrombopag is taken orally.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic soft tissue or bone sarcoma
* 18 years of age or older
* Adequate blood counts
* Adequate kidney and liver function
* At least 1 but no more than 3 prior systemic therapy regimens for this cancer
* Good performance status - able to carry out work of a light or sedentary nature

Exclusion Criteria:

* Pre-existing hear disease such as congestive heart failure, or arrhythmia known to increase the risk of thromboembolic events (blood clots)
* Blood clot in the last 6 months, known clotting problem or platelet disorder
* History of brain cancer

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Tolerated Eltrombopag Dose | 1 year
  Measured in milligrams (mg). The primary objective of the phase I study is to determine the recommended phase II dose. The maximum dose is the dose of which less than 2 of 6 patients experienced an unacceptable event/side effect
Efficacy | 20 weeks
  The primary outcome for the Phase II study is the proportion of subjects without grade 3 or 4 thrombocytopenia

CONTACTS AND LOCATIONS:
Overall Officials: Richard F Riedel, MD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States